CLINICAL TRIAL: NCT03190681
Title: Etude Comparative Monocentrique, Randomisée, En Cross-over, En Double Aveugle, Contre Placebo, De L'action Du Méthylphénidate Sur Les Paramètres Cognitifs De La Motivation
Brief Title: Motivation and Methylphenidate
Acronym: MBB_MPH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C13-08
Record Dates: First submitted 2017-05-31; First posted 2017-06-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Motivation; Apathy; Impulsive Behavior
MeSH Terms: conditions — Lethargy; Impulsive Behavior | interventions — Methylphenidate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methylphenidate then placebo (Experimental)
  Interventions: Drug: Ritalin 10Mg Tablet; Drug: Placebo Oral Tablet
- placebo then methylphenidate (Experimental)
  Interventions: Drug: Ritalin 10Mg Tablet; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ritalin 10Mg Tablet — oral ingestion of 3 tablets in a single-dose
Drug: Placebo Oral Tablet — oral ingestion of 3 tablets in a single-dose

SUMMARY:
The purpose of this study is to evaluate the impact of methylphenidate, a mixed dopaminergic and noradrenergic agent, onto the different components of motivation: decision-making, effort allocation and instrumental learning.

ELIGIBILITY:
Inclusion Criteria:

* weight>= 50kg and <=90kg
* free and informed consent
* social security affiliation
* no chronic illness
* no previous participation to a protocol wth similar tasks
* no special legal status (guardianship,trusteeship)
* no personnal or familial neurologic or psychiatric background
* no contraceptive device for a reproductive woman

Exclusion Criteria:

* inability to squeeze a handgrip
* smoking
* psychoactive substance consumption less than 3 weeks ago
* pregnant or breastfeeding woman
* hypersensitivity to methylphenidate
* hyperthyroidism
* cardiovascular or cerebrovascular disease
* respiratory, hepatic or renal failure
* glaucoma
* pheochromocytoma
* gluten intolerance or hypersensitivity
* galactosemia, glucose malabsorption syndrome, lactase deficit
* countraindicated meds (IMAO, IMAO-A, orhtosympathomimetics, alcaloids, linezolin, enzymatic inducers, psycho-active drugs)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
coefficient of sensitivity to reward | two hours after administration
  Parameter characterizing the influence of reward expectation/experience onto behavior for each individual.
  This parameter is estimated through the fit of computational models to behaviors recorded in a battery of motivational tasks (choice task, effort task, Learning task).

SECONDARY OUTCOMES:
coefficient of sensitivity to effort | two hours after administration
  Parameter characterizing the influence of effort expectation/experience onto behavior for each individual.
  This parameter is estimated through the fit of computational models to behaviors recorded in a battery of motivational tasks (choice task, effort task, Learning task).
coefficient of sensitivity to punishment | two hours after administration
  Parameter characterizing the influence of punishment expectation/experience onto behavior for each individual.
  This parameter is estimated through the fit of computational models to behaviors recorded in a battery of motivational tasks (choice task, effort task, Learning task).
coefficient of sensitivity to delay | two hours after administration
  Parameter characterizing the influence of delay expectation onto behavior for each individual.
  This parameter is estimated through the fit of computational models to behaviors recorded in a battery of motivational tasks (choice task, effort task, Learning task).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'investigation clinique, Institut du Cerveau et de la Moelle, Paris, France

IPD SHARING:
Plan to Share IPD: No